CLINICAL TRIAL: NCT06655727
Title: Evaluation of Dysphagia in Patients Diagnosed With Parkinson's Disease by Ultrasound: A Controlled Study
Brief Title: Evaluation of Dysphagia in Patients Diagnosed With Parkinson's Disease by Ultrasound
Status: Completed | Type: Observational
Sponsor: Beylikduzu State Hospital (Other)
Responsible Party: Principal Investigator, Busra Sirin, Principle Investigator, Beylikduzu State Hospital
Other Study IDs: BeylikduzuStateH5
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson disease group: Patients with Parkinson's disease
  Interventions: Diagnostic Test: Ultrasound evaluation
- Control group: Healthy volunteers
  Interventions: Diagnostic Test: Ultrasound evaluation

INTERVENTIONS:
Diagnostic Test: Ultrasound evaluation — No intervention

SUMMARY:
The primary aim of this study is to perform an ultrasonographic swallowing assessment in Parkinson's patients and healthy volunteers and compare the findings with those from clinical swallowing evaluations. The secondary aim is to examine the relationship between dysphagia and functional status.

DETAILED DESCRIPTION:
Thirty patients aged 40-80 years, diagnosed with idiopathic Parkinson's disease (Modified Hoehn-Yahr stage 1-3), and thirty healthy volunteers who either applied to the Physical Therapy and Rehabilitation outpatient clinic or received inpatient rehabilitation at Beylikdüzü State Hospital and Istanbul Physical Medicine and Rehabilitation Training and Research Hospital will be included in this study. At the start of the study, sociodemographic data of both patients and volunteers will be recorded. The Mini-Mental Test and the Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) will be used to evaluate the mental and functional status of the patients diagnosed with Parkinson's disease. After the clinical dysphagia evaluation, the EAT-10 questionnaire will be administered to the participants. Following this, an ultrasonographic swallowing assessment will be performed on the participants. The ultrasonographic measurements will include tongue thickness (cm), resting distance between the mandible and hyoid (cm), shortest distance between the mandible and hyoid (cm), hyoid displacement (cm), hyoid displacement percentage, tongue thickness (cm) (with 5ml of water), resting distance between the mandible and hyoid (cm) (with 5ml of water), shortest distance between the mandible and hyoid (cm) (with 5ml of water), hyoid displacement (cm) (with 5ml of water), and hyoid displacement percentage (%) (with 5ml of water).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease by a neurologist.
* Being in stages 1-3 according to the Modified Hoehn-Yahr Staging Scale.
* Scoring at least 24 on the Mini-Mental State Examination (MMSE).
* Not having received any therapy or treatment affecting swallowing, other than routine medication for Parkinson's disease.

Exclusion Criteria:

* Presence of head or neck cancer that could cause dysphagia.
* History of radiotherapy or surgery in the head and neck region.
* Diagnosis of vascular parkinsonism or stroke.
* Presence of cardiopulmonary disease that could affect swallowing or breathing.
* Having received voice or swallowing therapy in the last 6 months.
* Presence of a diagnosed psychiatric disorder.

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Parkinson's Disease and healthy controls
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-10-25 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
The EAT-10 (Eating Assessment Tool-10) | 0 day
  The EAT-10 (Eating Assessment Tool-10) is a validated self-administered questionnaire designed to assess symptoms of dysphagia (difficulty swallowing). It consists of 10 questions that evaluate the severity of swallowing difficulties, including issues related to eating, drinking, and managing saliva. Each item is rated on a 5-point scale, ranging from 0 (no problem) to 4 (severe problem). A total score of 3 or higher suggests the presence of clinically significant dysphagia, and it helps guide further diagnostic evaluation and management.
Unified Parkinson's Disease Rating Scale (UPDRS) | 0 day
  The UPDRS is a comprehensive tool used to evaluate the severity and progression of Parkinson's disease. It consists of multiple sections assessing motor and non-motor symptoms, helping clinicians understand the impact of the disease on daily functioning. The UPDRS is widely used in both clinical practice and research to monitor disease progression and treatment effects.
  In the MDS-UPDRS, higher scores indicate more severe Parkinson's disease symptoms. Each item is rated from 0 (normal) to 4 (severe), with the total score reflecting the overall disease severity. A higher total score means worse motor and non-motor symptoms, indicating greater impairment and reduced quality of life. Lower scores suggest milder symptoms and better functional status.

SECONDARY OUTCOMES:
Tongue Thickness | 0 day
  Tongue thickness refers to the measurement of the width or thickness of the tongue in centimeters. This parameter is evaluated using ultrasound to assess the muscle mass and structural integrity of the tongue, which plays a critical role in swallowing function. In conditions like dysphagia, reduced tongue thickness may indicate weakened tongue muscles, contributing to swallowing difficulties.
Distance Between the Hyoid and Mandible | 0 day
  This is the measurement of the space between the hyoid bone and the mandible (lower jaw) while the individual is at rest or during swallowing. It is typically measured in centimeters and can provide insights into the positioning and movement of structures involved in swallowing. An abnormal distance between these structures may indicate dysfunction in the swallowing mechanism.
Hyoid Displacement Distance: | 0 day
  The hyoid bone plays a key role in the swallowing process by facilitating the elevation and forward movement of the larynx. Insufficient hyoid displacement can lead to impaired swallowing function, as it affects the coordination of muscles involved in the swallow. The measurement of this displacement helps assess the efficiency and safety of the swallowing mechanism.

CONTACTS AND LOCATIONS:
Locations (1):
- Beylikdüzü State Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No